CLINICAL TRIAL: NCT06456892
Title: Phase I/II Clinical Study on the Safety and Effectiveness of Pucotenlimab Combined With Standard Chemotherapy Regimen as Neoadjuvant Therapy for Children and Adolescents With Intermediate/High-Risk Rhabdomyosarcoma
Brief Title: Effectiveness of Pucotenlimab Combined With Standard Chemotherapy Regimen
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Chief of Department of pediatric oncology, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pucotenlimab-01
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Rhabdomyosarcoma; Pediatric Cancer
MeSH Terms: conditions — Rhabdomyosarcoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pucotenlimab Combined with Standard Chemotherapy Regimen (Experimental): In phase I, it focuses on safety, tolerability, and pharmacokinetics using a "3+3" dose escalation design with three dose groups: 1 mg/kg, 3 mg/kg, and 6 mg/kg. The drug will be administered in combination with the standard regimen for intermediate/high-risk rhabdomyosarcoma once every three weeks (Q3W).
  In phase II, after establishing the recommended Phase II dose (RP2D), ll subjects will receive Pucotenlimab combined with the standard regimen for intermediate/high-risk rhabdomyosarcoma for 2-4 cycles of neoadjuvant therapy every 3 weeks (Q3W), followed by surgery.
  The standard regimen for intermidiate/high-risk rhabdomyosarcoma refer to the SYSUCC-RMS-2017 in China.
  Interventions: Drug: Pucotenlimab

INTERVENTIONS:
Drug: Pucotenlimab — Pucotenlimab Combined with Standard Chemotherapy Regimen

SUMMARY:
This study comprises both Phase I and Phase II research. This phase focuses on safety, tolerability, and pharmacokinetics using a "3+3" dose escalation design with three dose groups: 1 mg/kg, 3 mg/kg, and 6 mg/kg. The drug will be administered in combination with the standard regimen for intermediate/high-risk rhabdomyosarcoma once every three weeks (Q3W). In phase II study, all subjects will receive Pucotenlimab combined with the standard regimen for intermediate/high-risk rhabdomyosarcoma for 2-4 cycles of neoadjuvant therapy every 3 weeks (Q3W), followed by surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1-18 years old;
2. ECOG PS score: 0-1 points;
3. Pathologically confirmed newly diagnosed children or adolescents with intermediate to high-risk rhabdomyosarcoma;
4. Patients evaluated by surgery as having a high degree of difficulty;
5. Must have at least one measurable lesion defined by RECIST or WHO criteria;
6. Expected survival time ≥ 6 months;
7. Cardiac function:

   1. Echocardiography shows LVEF ≥ 50%;
   2. EKG indicates no evidence of myocardial ischemia;
   3. No history of arrhythmia requiring pharmacological intervention before enrollment;
8. No history of severe immune-related adverse events (CTCAE V4.03 G3 or G4);
9. For patients with known non-involvement of the bone marrow (BM):

   1. Absolute neutrophil count (ANC) ≥ 1.0 × 109/L;
   2. Platelet count ≥ 100.0 × 109/L;
   3. Hemoglobin ≥ 90 g/L;
10. Liver and kidney functions need to meet the following criteria:

    1. Total bilirubin (conjugated + unconjugated) ≤ 2.5 × upper limit of normal (ULN) corresponding to age, patients with confirmed Gilbert's syndrome may be enrolled based on the investigator's discretion;
    2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN;
    3. Estimated glomerular filtration rate ≥ 30 mL/min/1.73 m2 or serum creatinine (Cr) ≤ 1.5 × ULN;
11. Able to comply with outpatient treatment, laboratory monitoring, and necessary clinical visits during the study;
12. The parents/guardians of the child or adolescent participants have the ability to understand, consent to, and sign the informed consent form (ICF) and applicable child consent forms before initiating any protocol-related procedures; the participants have the ability to express their consent (if applicable) with the consent of their parents/guardians.

Exclusion Criteria:

1. Received anti-PD-1 or anti-PD-L1 monoclonal antibodies or targeted drugs related to these pathways;
2. Received chemotherapy, radiotherapy, or other treatments;
3. Previous surgical treatment (excluding biopsy);
4. Known allergy to PD-1 monoclonal antibodies or any of their excipients; known history of allergic diseases or severe allergies;
5. Having other malignant tumor diseases besides the tumor being treated in this study, excluding: malignant tumors that have been cured and have not recurred within 3 years before enrollment, completely resected basal cell and squamous cell skin cancers, completely resected carcinoma in situ of any type;
6. Active central nervous system metastases (whether treated or not), including symptomatic brain metastases, meningeal metastases, or spinal cord compression, etc. Excluding: asymptomatic brain metastases without progression within at least 4 weeks after radiotherapy and/or without neurological symptoms or signs after surgical resection, without the need for dexamethasone or mannitol treatment.
7. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
8. Previous treatment toxicity still > Grade 1 (CTCAE V4.03 criteria), excluding alopecia and neurotoxicity;
9. History of mental disorders;
10. History of drug abuse or substance abuse upon inquiry;
11. History of idiopathic pulmonary fibrosis or idiopathic pneumonitis;
12. Comorbidities requiring immunosuppressive drug treatment, or comorbidities requiring systemic or local use of corticosteroids at immunosuppressive doses (prednisone > 10 mg/day or equivalent doses of similar drugs).
13. History of autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, etc. Excluding: Type I diabetes, hypothyroidism controllable only through hormone replacement therapy, dermatological diseases that do not require systemic treatment (such as vitiligo, psoriasis), controlled celiac disease, or diseases that are not expected to recur without external stimuli;
14. Previous or current active tuberculosis infection;
15. Active infections requiring systemic treatment;
16. Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg) or pulmonary hypertension or unstable angina pectoris; myocardial infarction or bypass surgery, stenting within 6 months before administration; history of chronic heart failure satisfying New York Heart Association (NYHA) Class 3-4; clinically significant valvular heart disease; severe arrhythmias requiring treatment (excluding atrial fibrillation, paroxysmal supraventricular tachycardia), including QTc interval ≥ 450 ms for males and ≥ 470 ms for females (calculated using the Fridericia formula); cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months before administration;
17. Concurrent severe medical conditions, including but not limited to: uncontrolled diabetes, active peptic ulcer, active bleeding, etc.;
18. Positive Anti-HIV, TP-Ab, HCV-Ab; HBV-Ag positive with HBV DNA copy number > upper limit of normal value of the testing unit;
19. Abnormal thyroid function test results (FT3, FT4, T3, T4);
20. Expected to receive live or attenuated vaccines within 4 weeks before administration, during treatment, or within 5 months after the last dose;
21. Participated in another clinical trial and received experimental drug treatment within 30 days before administration;

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
DLT | within 28 days of the dose escalation phase.
  dose-limiting toxicity
pCR | from treatment of pucotenlimab to the surgery
  pathological complete response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No